CLINICAL TRIAL: NCT00365157
Title: A Phase I/II Study of E7389 Halichondrin B Analog (NSC # 707389) in Metastatic Urothelial Tract Cancer and Renal Insufficiency
Brief Title: Eribulin Mesylate in Treating Patients With Locally Advanced or Metastatic Cancer of the Urothelium and Kidney Dysfunction
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00170; NCI-2009-00170 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000492014; PHII-75; 7435 (Other: City of Hope Comprehensive Cancer Center); 7435 (Other: CTEP); N01CM00038 (NIH); N01CM00071 (NIH); N01CM62201 (NIH); N01CM62209 (NIH); P30CA033572 (NIH); U01CA062505 (NIH); UM1CA186705 (NIH); UM1CA186717 (NIH)
Record Dates: First submitted 2006-08-16; First posted 2006-08-17 (Estimated); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Advanced Urothelial Carcinoma; Locally Advanced Urothelial Carcinoma; Metastatic Urothelial Carcinoma; Recurrent Urothelial Carcinoma; Stage III Bladder Urothelial Carcinoma AJCC v6 and v7; Stage IV Bladder Urothelial Carcinoma AJCC v7; Unresectable Urothelial Carcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — eribulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (eribulin mesylate) (Experimental): Patients receive eribulin mesylate IV over 1-2 minutes on days 1 and 8. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Eribulin Mesylate; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study

INTERVENTIONS:
Drug: Eribulin Mesylate — Given IV
  Other Names: B1939 Mesylate; E7389; ER-086526 Mesylate; Halaven; Halichondrin B Analog
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies

SUMMARY:
This phase I/II trial studies the effect of eribulin mesylate and to see how well it works in treating patients with cancer of the urothelium that has spread to nearby tissue (locally advanced) or to other places in the body (metastatic)and kidney dysfunction. Drugs used in chemotherapy, such as eribulin mesylate, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Chemotherapy drugs may have different effects in patients who have changes in their kidney function.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To establish whether eribulin mesylate (E7389) can be given safely to patients with moderate and severe renal dysfunction at 1.4 mg/m^2/week (the maximum tolerated dose [MTD] previously defined for patients with normal renal function) on days 1 and 8 of a 21-day cycle. (Phase I) II. To characterize the pharmacokinetic (PK) profile of E7389 in patients with moderate and severe renal dysfunction. (Phase I) III. To determine the response rate of patients with advanced urothelial carcinomas to E7389 in the first-line setting. (Phase II) IV. To determine the 6-month, progression-free survival and overall survival of patients with advanced urothelial carcinomas treated with E7389. (Phase II) V. To document the toxicity associated with the administration of E7389 to patients with advanced urothelial carcinoma patients and varying degrees of renal dysfunction. (Phase II) VI. To determine the response rate of patients with advanced urothelial carcinomas to E7389 in the setting of progression after prior platinum-based chemotherapy for advanced or recurrent disease, in two cohorts: tubulin-inhibitor treated or tubulin-inhibitor naive. (tubulin inhibitors in common use for urothelial cancer include paclitaxel, docetaxel and vinblastine). (Phase II) (per Amendment 6) VII. To determine the 6-month progression-free survival and overall survival of patients with advanced urothelial carcinomas treated with E7389 after platinum-based therapy for recurrent or advanced disease. (Phase II) (per Amendment 6) VIII. To document the toxicity associated with the administration of E7389 to patients with advanced urothelial carcinoma patients in the second line and later setting. (Phase II) (per Amendment 6) IX. To compare men and women with advanced bladder cancer treated with E7389 with respect to toxicity of E7389 as classified by Common Terminology Criteria for Adverse Events (CTCAE) version (v)4 for (i) all hematologic toxicities, (ii) all non- hematologic toxicities, and (iii) the most frequently observed toxicities (neutropenia, anemia, leucopenia, infection). (Enrollment to additional females) (per Amendment 11) X. To compare men and women with advanced bladder cancer treated with E7389 with respect to response to E7389 as evidenced by (i) disease control rate (DCR) defined as stable disease (SD)+partial response (PR)+complete response (CR) at 12 weeks, (ii) progression-free survival (PFS), and (iii) overall survival (OS). (Enrollment to additional females) (per Amendment 11) XI. To compare men and women with advanced bladder cancer treated with E7389 with respect to pharmacokinetics of E7389. (Enrollment to additional females) (per Amendment 11) XII. To compare men and women with advanced bladder cancer treated with E7389 with respect to tumoral expression of genes involved in the mechanism of action of E7389, including tubulin isotypes, microtubule-associated protein 4 (MAP4), and stathmin. (Enrollment to additional females) (per Amendment 11)

OUTLINE:

Patients receive eribulin mesylate intravenously (IV) over 1-2 minutes on days 1 and 8. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up monthly for 12 months and then every 3 months for up to 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have locally advanced or metastatic urothelial cancer that is not amenable to surgical treatment
* Patients must have histologically or cytologically confirmed urothelial tract carcinoma
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >= 20 mm with conventional techniques or as >= 10 mm with spiral computed tomography (CT) scan
* All patients may have received up to two prior lines of chemotherapy for recurrent/advanced disease
* Patients must have received at least one platinum-based chemotherapy for recurrent/advanced disease; recurrent disease is defined as having recurred after definitive therapy and advanced disease is defined as T4 and/or N2 and/or M1; in addition, for completion of Cohort #2, patients must also have received a tubulin inhibitor as part of their therapy for urothelial cancer; for purposes of this evaluation, treatment with chemotherapy regimens where carboplatin or similar is substituted for cisplatin or where a taxane is added or removed will be considered the same regimen; tubulin inhibitors in common use include paclitaxel, docetaxel, and vinblastine; the exception to this requirement applies to women
* Women with and without prior therapy are also eligible; priority will be given to those who consent to participating in the pharmacokinetic studies
* Life expectancy of greater than 6 months
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2 and Karnofsky >= 60%
* Absolute neutrophil count >= 1,000/mcL
* Platelets >= 100,000/mcL
* Hemoglobin >= 9 g/dL
* Total bilirubin =< 1.5 institutional upper limit of normal (IULN)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 X IULN
* Patients must have either (a) normal kidney function (i.e. creatinine =< 1.5 X upper limit of normal [ULN] OR calculated creatinine clearance >= 60 mL/min by the modified Cockcroft and Gault Formula OR a creatinine clearance >= 60 mL/min obtained from a 24-hour urine collection) or (b) moderate or severe renal dysfunction (i.e. creatinine clearance < 60 mL/min and >= 20 mL/min)
* Patients with symptomatic uremia, uncontrolled edema or unstable serum electrolytes should not enter the trial until such time as they have been stabilized - such patients should be discussed with the principal investigator
* Eligibility of patients receiving any medications or substances known to affect or with the potential to affect the activity or pharmacokinetics of E7389 Halichondrin analog will be determined following review of their case by the principal investigator
* The effects of E7389 Halichondrin analog on the developing human fetus at the recommended therapeutic dose are unknown; for this reason and because tubulin inhibitors are known to be teratogenic, women and men of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Patients must have the ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients may not be receiving any other investigational agents
* Patients with brain metastasis that are unstable (i.e. presenting with neurologic symptoms that progress or require increasing doses of steroids within a 4-week period) or are untreated (i.e. not radiated) should be excluded
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because E7389 Halichondrin analog is tubulin inhibitor agent with the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with E7389 Halichondrin analog, breastfeeding should be discontinued if the mother is treated with E7389
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with E7389 Halichondrin analog; HIV-positive patients with CD4+ =< 500/mm3 are ineligible because they are at increased risk of lethal infections when treated with marrow-suppressive therapy; appropriate studies will be undertaken in this group of patients when indicated
* Prior therapy with E7389 Halichondrin analog (eribulin)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2006-10-23 (Actual); Primary Completion 2025-07-09 (Actual); Study Completion 2026-07-09 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) and recommended phase II dose (RP2D) of eribulin mesylate for patients who have received a tubulin-inhibitor for the recurrent/advanced disease (Phase I) | 21 days
  MTD and RP2D will be graded according to Common Terminology Criteria for Adverse (CTCAE) version 5.0.
MTD and RP2D of eribulin mesylate for patients who have not received a tubulin-inhibitor for the recurrent/advanced disease (Phase I) | 21 days
  MTD and RP2D will be graded according to CTCAE version 5.0.
Overall response rate | Up to 6 months
  Calculated as the ratio of the number of eligible patients who experienced a confirmed complete response (CR) or partial response (PR) by Response Evaluation Criteria in Solid Tumors version 1.1 (Phase II). 95% confidence intervals will be constructed.

SECONDARY OUTCOMES:
Progression-free survival (Phase II) | From the start of treatment on day 1 until progression, death, or the start of another treatment, assessed at 6 months
  Summarized with Kaplan-Meier plots and confidence intervals. The Cox proportional hazards model will be used to compare males and females, adjusting for the pharmacokinetic (PK) variables as well as age, renal status, and prior therapy.
Progression-free survival (Phase II) | From the start of treatment on day 1 until progression, death, or the start of another treatment, assessed up to 12 months
  Summarized with Kaplan-Meier plots and confidence intervals. The Cox proportional hazards model will be used to compare males and females, adjusting for the PK variables as well as age, renal status, and prior therapy.
Overall survival (Phase II) | From the start of treatment on day 1 until progression, death, or the start of another treatment, assessed up to 12 months
  Summarized with Kaplan-Meier plots and confidence intervals. The Cox proportional hazards model will be used to compare males and females, adjusting for the PK variables as well as age, renal status, and prior therapy.
Incidence of adverse events | Up to 24 months
  Graded according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. All observed toxicities will be summarized in terms of type (organ affected or laboratory determination such as absolute neutrophil count), severity (by the CTCAE version 5.0), and time of onset (i.e. course of treatment). Tables will be created to summarize these toxicities and side effects, overall, by course, by renal insufficiency status, and by prior exposure to tubulin-inhibitors.

OTHER OUTCOMES:
Pharmacokinetic parameters for eribulin mesylate | At baseline; at 5, 10, 15, and 30 minutes; and at 1, 2, 4, 6, 8, 12, and 24 hours on day 1 of course 1 and at end of days 2-4 and 8 of course 1
  Analyzed using compartmental and non-compartmental models. max concentration, systemic clearance, renal clearance, volume of distribution, half life, and area under the curve tabulated overall, and by prior exposure to tubulin-inhibitors, with summary statistics (means and standard deviations, or medians and ranges) and displayed with box-plots; the relationship between the PK parameters and indices of renal function (e.g. serum creatinine and creatinine clearance) will be examined using scatterplots and correlations.
Expression levels of the tubulin isotypes | Baseline
  For each of the tubulin isotypes, the distribution of the expression levels will be summarized with plots and standard statistical summary numbers; prior to analysis, the expression levels may be transformed to render the distributions more compatible with the assumptions of normal distribution. The association between the expression levels and response will be summarized with means and standard deviations and confidence intervals (or medians and ranges) and displayed with box-plots.
Disease control rate (complete response [CR] + partial response [PR] + stable disease [SD]) | 12 weeks
  Logistic regression will be used to compare males and females, adjusting for the PK variables as well as age, renal status, and prior therapy.

CONTACTS AND LOCATIONS:
Overall Officials: David I Quinn, Principal Investigator — City of Hope Comprehensive Cancer Center
Locations (26):
- United States (26):
  - Tower Cancer Research Foundation, Beverly Hills, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - City of Hope Antelope Valley, Lancaster, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Veterans Administration Hospital - Martinez, Martinez, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - City of Hope South Pasadena, South Pasadena, California
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Duly Health and Care Joliet, Joliet, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Fort Wayne Medical Oncology and Hematology Inc-Parkview, Fort Wayne, Indiana
  - Community Howard Regional Health, Kokomo, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Oncology Care Associates PLLC, Saint Joseph, Michigan
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Medical College of Wisconsin, Milwaukee, Wisconsin